CLINICAL TRIAL: NCT04091789
Title: A Controlled-Dose Study Using Cannabinoid Combinations in a Rapidly Dissolvable Sublingual Tablet for the Treatment of Dysmenorrhea and Associated Pain Symptoms
Brief Title: Sublingual Tablets With Cannabinoid Combinations for the Treatment of Dysmenorrhea
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pure Green (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PG-19-003
Record Dates: First submitted 2019-09-13; First posted 2019-09-17 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Dysmenorrhea; Headache, Migraine; Fatigue; Nausea; Mood Disturbance
Keywords: Pain Associated with Dysmenorrhea; CBD; Cannabidiol
MeSH Terms: conditions — Dysmenorrhea; Migraine Disorders; Fatigue; Nausea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test Article (Experimental): Subjects will take Pure Femme sublingual tablets as directed, one tablet 2 days before, one tablet 1 day before, and then up to 3 tablets per day for 3 days (72 hours) during menstruation.
  Interventions: Drug: Pure Femme Tablets

INTERVENTIONS:
Drug: Pure Femme Tablets — A sublingual tablet containing 30 mg of cannabidiol (CBD), 1 mg tetrahydrocannabinol (THC), 97 mg palmitoylethanolamide (PEA), and a 0.2 mg combination of myrcene, beta-caryophyllene, humulene, linalool, and limonene and peppermint oil.

SUMMARY:
Sublingual Tablets With Cannabinoid Combinations for the Treatment of Dysmenorrhea

ELIGIBILITY:
Inclusion Criteria:

1. Subject is female and at least 21 years of age;
2. Subject has a regular, predictable menstrual cycle ranging in length from 21-35 days;
3. Subject has a diagnosis of primary dysmenorrhea with an average pain scale score of 5 or greater;
4. Subject is willing to provide her informed consent via DocuSign to participate in the study as stated in the informed consent document.
5. Subject knows how to use and is willing to use a smart phone app to record information.

Exclusion Criteria:

1. Subject is pregnant or lactating;
2. Subject has an allergy to cannabis (marijuana), the Cannabaceae plant family (e.g., hemp, hops), PEA, terpenes, citrus, or lavender, peppermint;
3. Subject has a known allergy to active or inert ingredients of Pure Femme tablets;
4. Subject is taking a concomitant medication or treatment that would complicate use or interpretation of the study drug's effects (examples include: Cannabis or any cannabinoid products including CBD and THC; Any drug or herbal product that influences the endocannabinoid system (ECS));
5. Subject has a history of endometriosis, pelvic inflammatory disease, adenomyosis, leiomyomata, or chronic pelvic pain;
6. Subject has a history of migraines, tension headaches, or cluster headaches not associated with menstruation or is currently taking medication for headache treatment or prevention (e.g., tricyclic antidepressants, beta-blockers, anticonvulsants, triptans);
7. Subject is currently using any of the following medications or classes of medication routinely: opioids, anti-emetics, acetaminophen, NSAIDS, ergotamines, triptans, or, glucocorticoids;
8. Subject has shortness of breath associated with allergies;
9. Subject has uncontrolled asthma;
10. Subject has a fever and/or productive cough.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Qualifying subjects must have regular, predictable menstrual cycles that range in length between 21-35 days.
Enrollment: 30 (Estimated)
Dates: Start 2019-09 (Estimated); Primary Completion 2020-03 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Impact of Pure Green tablet on menstrual pain as measured by a pain scale score | Two Months
  The study objective is to examine the impact on Pure Green tablet on menstrual related pain. Patients will self report their pain scale score using 0-10 scale where 0 is no pain and 10 is the worst pain ever.

SECONDARY OUTCOMES:
The impact of Pure Green tablets will be measured by the WHO QOL questionnaire comparing pre and post dosing responses. | Two Months
  Subjective quality of life during menses will be measured by using the World Health Organization's Quality of Life (QOL) questionnaire. Patients will be asked a rating scale 1-5 where 1 is not at all and 5 is an extreme amount of elements such as health, enjoyment, happiness, concentration, energy levels, at the beginning and end of their menstrual cycle and results will be compared.
The impact of Pure Green tablets will be compared to patient's usual treatment of mentrual pain. | Two Months
  Patients be asked which medications and doses are usually taken to treat menstrual related symptoms. During the trial, patients will document any additional medications taken and if so, the amount of the medications needed beyond the trial drug in order to treat their menstrual related symptoms. The results will be compared to what they originally documented as their usual therapeutic treatment.
Impact of Pure Green tablets on mood disturbance as measured by the Steiner PMTS questionnaire. | Two Months
  The Steiner rating scale will be used to evaluate mood disturbances during menses and the impact of Pure Green tablets on mood disturbances during menses. A scale of 0-4 where 0 is the absence of the mood and 4 is severe will be used to examine elements such as irritability, tension, dysphoria, fatiguability, coordination, cognitive functioning, eating habits, and social impairment. The results will be compared with a self-reported pre-study accounting of usual mood during menses.
Evaluate the impact of Pure Green tablets on menstrual related headache or migraine as evaluated by a questionnaire | Two Months
  Patients will be given a headache specific questionnaire before and after the trial to assess the impact of Pure Green tablets on menstrual related migraine or headache. The questionnaire is comprised of 4 yes or no questions asking about headache and or migraine related to menstruation. The results will be compared with the pre-study self reporting of headache or migraine during menstruation.

CONTACTS AND LOCATIONS:
Overall Officials: Debra Kimless, M.D., Principal Investigator — Pure Green
Locations (1):
- Dr. Nakadar's Office, Sterling Heights, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baker FC, Driver HS, Rogers GG, Paiker J, Mitchell D. High nocturnal body temperatures and disturbed sleep in women with primary dysmenorrhea. Am J Physiol. 1999 Dec;277(6):E1013-21. doi: 10.1152/ajpendo.1999.277.6.E1013. PMID 10600789
- [Background] Chantler I, Mitchell D, Fuller A. Actigraphy quantifies reduced voluntary physical activity in women with primary dysmenorrhea. J Pain. 2009 Jan;10(1):38-46. doi: 10.1016/j.jpain.2008.07.002. Epub 2008 Aug 23. PMID 18722817
- [Background] Dorn LD, Negriff S, Huang B, Pabst S, Hillman J, Braverman P, Susman EJ. Menstrual symptoms in adolescent girls: association with smoking, depressive symptoms, and anxiety. J Adolesc Health. 2009 Mar;44(3):237-43. doi: 10.1016/j.jadohealth.2008.07.018. Epub 2008 Oct 29. PMID 19237109
- [Background] Harel Z. Dysmenorrhea in adolescents and young adults: etiology and management. J Pediatr Adolesc Gynecol. 2006 Dec;19(6):363-71. doi: 10.1016/j.jpag.2006.09.001. PMID 17174824
- [Background] Iacovides S, Avidon I, Bentley A, Baker FC. Reduced quality of life when experiencing menstrual pain in women with primary dysmenorrhea. Acta Obstet Gynecol Scand. 2014 Feb;93(2):213-7. doi: 10.1111/aogs.12287. Epub 2013 Nov 25. PMID 24266425
- [Background] Jamieson DJ, Steege JF. The prevalence of dysmenorrhea, dyspareunia, pelvic pain, and irritable bowel syndrome in primary care practices. Obstet Gynecol. 1996 Jan;87(1):55-8. doi: 10.1016/0029-7844(95)00360-6. PMID 8532266
- [Background] Latthe PM, Champaneria R. Dysmenorrhoea. BMJ Clin Evid. 2014 Oct 21;2014:0813. PMID 25338194
- [Background] Latthe P, Latthe M, Say L, Gulmezoglu M, Khan KS. WHO systematic review of prevalence of chronic pelvic pain: a neglected reproductive health morbidity. BMC Public Health. 2006 Jul 6;6:177. doi: 10.1186/1471-2458-6-177. PMID 16824213
- [Background] Latthe P, Mignini L, Gray R, Hills R, Khan K. Factors predisposing women to chronic pelvic pain: systematic review. BMJ. 2006 Apr 1;332(7544):749-55. doi: 10.1136/bmj.38748.697465.55. Epub 2006 Feb 16. PMID 16484239
- [Background] Lefebvre G, Pinsonneault O, Antao V, Black A, Burnett M, Feldman K, Lea R, Robert M; SOGC. Primary dysmenorrhea consensus guideline. J Obstet Gynaecol Can. 2005 Dec;27(12):1117-46. doi: 10.1016/s1701-2163(16)30395-4. English, French. PMID 16524531
- [Background] Marjoribanks J, Proctor M, Farquhar C, Derks RS. Nonsteroidal anti-inflammatory drugs for dysmenorrhoea. Cochrane Database Syst Rev. 2010 Jan 20;(1):CD001751. doi: 10.1002/14651858.CD001751.pub2. PMID 20091521
- [Background] Proctor M, Farquhar C. Diagnosis and management of dysmenorrhoea. BMJ. 2006 May 13;332(7550):1134-8. doi: 10.1136/bmj.332.7550.1134. No abstract available. PMID 16690671
- [Background] Stegeman BH, de Bastos M, Rosendaal FR, van Hylckama Vlieg A, Helmerhorst FM, Stijnen T, Dekkers OM. Different combined oral contraceptives and the risk of venous thrombosis: systematic review and network meta-analysis. BMJ. 2013 Sep 12;347:f5298. doi: 10.1136/bmj.f5298. PMID 24030561
- [Background] Wang T, Collet JP, Shapiro S, Ware MA. Adverse effects of medical cannabinoids: a systematic review. CMAJ. 2008 Jun 17;178(13):1669-78. doi: 10.1503/cmaj.071178. PMID 18559804
- [Background] Zannoni L, Giorgi M, Spagnolo E, Montanari G, Villa G, Seracchioli R. Dysmenorrhea, absenteeism from school, and symptoms suspicious for endometriosis in adolescents. J Pediatr Adolesc Gynecol. 2014 Oct;27(5):258-65. doi: 10.1016/j.jpag.2013.11.008. Epub 2014 Apr 18. PMID 24746919